CLINICAL TRIAL: NCT05474651
Title: Influencing Factors and Trigger Mechanism of Relapse in Expectant Fathers Who Quit Smoking: An Exploratory Sequential Mixed Methods Study.
Brief Title: Influencing Factors and Trigger Mechanism of Relapse in Expectant Fathers Who Quit Smoking
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, A.P., Sun Yat-sen University
Other Study IDs: wjn-relapse（father）-2022.07
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation
Keywords: Expectant fathers; Smoking relapse; Mix-method study; Paternal Behavior
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed expectant fathers who quit smoking: Participants who met the inclusion criteria below will be invited to fill in the questionnaires set, part of them will be invited to attend a semi-structured interview(optional).
  1. Males ≥18 years old;
  2. The wife has given birth, the newborn is live, and the number of days of birth is less than or equal to 28 days;
  3. Self-reported smoking at least 1 cigarette per day on average for at least 1 month in the past 1 year;
  4. Self-reported that they had quit smoking during their wife's pregnancy on purpose, and maintained it for at least 24 hours;
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information sheet, characteristics of smoking sheet, the Fagerstrom Test of Nicotine Dependence,Smoking Self-efficacy Questionnaire, Cigarette Withdrawal Scale, smoking hazard questionnaire, motivation to quit smoking sheet, ability to quit smoking sheet, alcohol consumption, International Physical Activity Questionnaire.

SUMMARY:
The purpose of this study is to describe the relapse rate and characteristics of expectant fathers who quit smoking during their wives' pregnancy, to explore the influencing factors and triggering mechanisms,and describe their experience.

DETAILED DESCRIPTION:
Participants will be invited to recall their smoking status and experience during their wife's pregnancy (all participants and required to complete the questionnaire, and some of them will be invited to participate in semi-structured interviews).

In the quantitative study,participants need to finish the questionnaire,which includes the demographic information sheet, characteristics of smoking sheet, history of smoking cessation sheet, smoking hazard questionnaire, motivation to quit smoking sheet, ability to quit smoking sheet, alcohol consumption, exercise.

In the qualitative study,participants need to participate in semi-structured interview.The interview begins with "Have you tried smoking cessation before? Why? What is the result", and explores in-depth analysis based on the participants' answers.

ELIGIBILITY:
Inclusion Criteria:

* (1) All participants should be aged 18 or above;
* (2) The newborn of the participant is alive, and the number of days of birth is ≤28 days;
* (3) All participants should have actively quit smoking during his wife's pregnancy, and maintained it for at least 24 hours;
* (4) All participants should be smoking at least 1 cigarette per day on average for at least 1 month in the past 1 year;
* (5) All participants should be able to communicate in Mandarin (including reading Chinese).

Exclusion Criteria:

* All participants who meet the above criteria but are currently involved in other smoking cessation programs or the pilot study and/or mentally or physically unfit for communication will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The participant eligibility is based on both biological and self-representation of gender identity, smokers who is male biologically and also reported as a male will be eligible in this study
Study Population: The investigators will be admitted to the maternity ward of the partner hospital.
  Convenience sampling will be conducted, and expectant fathers who meet the criteria will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Smoking relapse rate | Baseline
  A true or false sheet in the questionnaire.

SECONDARY OUTCOMES:
Quality of relationship | Baseline
  The quality of relationship will be assessed by using the Relationship Satisfaction scale.It includes five items and a six-point response format was used, ranging from 'strongly disagree' to 'strongly agree'.
Withdrawal symptoms | Baseline
  The Cigarette Withdrawal Scale(CWS) is composed of 21 items, including four measuring depression-anxiety, four measuring craving, four measuring irritability-impatience, three measuring concentration difficulties, three measuring appetite-weight gain, and three measuring insomnia. The items were scored using a 5-point Likert-type scale (agree/disagree).
Self-efficacy level | Baseline
  Self-efficacy of participants against tobacco will be assessed by using by the Smoking Self-Efficacy Questionnaire(SEQ-12). The SEQ-12 is categorized into two subscales, namely internal stimuli (6 items) and external stimuli (6 items), with total possible scores ranging from 6 to 30 for both internal stimuli and external stimuli. Higher scores of the SEQ-12 on both subscales indicate greater selfefficacy to refrain from smoking.
Dependence of nicotine | Baseline
  The level of nicotine dependence of the participants will be measured by the Fagerstrom Test of Nicotine Dependence (FTND) scale. The FTND is a standard instrument for assessing the intensity of physical addiction to nicotine.The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerstrom score, the more intense is the patient's physical dependence on nicotine.
Self-awareness of the hazard of smoking | Baseline
  The self-awareness of the hazard of smoking among the participants will be measured by a self-designed smoking hazard questionnaire list. The 20-items questionnaire is developed according to the literature review content, focusing on the impact of smoking hazard on maternal and neonate health.Participants were asked to answer whether the knowledge about tobacco harm contained in the entry is correct: yes, no, or don't know (about 20% interference items).The higher the total score,the better the mastery of self-awareness of the hazard of smoking.
Smoking rationalization | Baseline
  The smoking rationalization will be measured by a 26-item scale within six dimensions (smoking functional beliefs, risk generalization beliefs, social acceptability beliefs, safe smoking beliefs, self-exempting beliefs, and quitting is harmful beliefs). Each item used a 5-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neither disagree nor agree, 4 = agree, 5 = strongly agree, higher scores represent higher levels of rationalization).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.